CLINICAL TRIAL: NCT06044181
Title: Long Term Management of Peripheral Avascular Retina in Retinopathy of Prematurity Evaluated by Fundus Fluorescein Angiography.
Brief Title: Peripheral Avascular Retina in Retinopathy of Prematurity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alyaa mohamed yousef ahmed elkabsh, principle investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Avascular Retina in ROP
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-09

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral avascular retina of ROP with no leakage. (No Intervention): If there is no active leakage detected by FFA, patients would be observed. The follow-up period: FFA will be done at the age of 18 months we will repeat FFA every 6 months and fundus examination with color photography every 3 months till the age of 3 years of children.
- Peripheral avascular retina of ROP with active leakage. (Active Comparator): If there is evidence of active leakage by FFA The confluent laser burns will be applied to the entire avascular retina from the ridge to the ora serrata for 360 through the transpupillary route.
  Interventions: Procedure: Diode laser photocoagulation.

INTERVENTIONS:
Procedure: Diode laser photocoagulation. — If there is evidence of active leakage by FFA The confluent laser burns will be applied to the entire avascular retina from the ridge to the ora serrata for 360 through the transpupillary route. The laser settings used are: power 250-400 mW and duration of 200-400 ms for 810 nm DLPC.
  Arms: Peripheral avascular retina of ROP with active leakage.

SUMMARY:
Retinopathy of prematurity (ROP) is a widely known retinal vascular disorder in preterm infants and a leading cause of visual disability or blindness in children. Advances in antenatal care have resulted in an increase in the survival rate of infants with extremely low birth weight (BW). Approximately 90% of infants who develop ROP do so by a postmenstrual age of 46.3 weeks. In certain patients with or without treatment, the retina may fail to fully vascularize or may develop vascular abnormalities, thus demonstrating persistent avascular retina (PAR) or anomalous vessel findings at the periphery. Because of the advent of technologies such as ultrawide-field fluorescein angiography (UWFFA) persistent vascular abnormalities can be detected more readily and investigated.

DETAILED DESCRIPTION:
The natural history of peripheral nonperfusion and vascular abnormalities, which persist beyond the acute phase of ROP, remains poorly understood. Although patients with a history of type I ROP (treatment requiring ROP) are more likely to exhibit abnormal foveal development and poor vision, a discrepancy still exists between the structural and functional findings of vascular abnormalities in the long term. For instance, circumferential atypical vessels are detected in patients with spontaneously regressed ROP and favorable vision. Additionally, persistent retinal vascular abnormalities may not necessarily predict adverse functional outcomes. The significance of such vessel anomalies and whether they persist or not remain uncertain. The physiologic avascular retina of children of age < 13 years usually extends ≤ 1.5 DD temporally or ≤ 1.0 DD nasally from the ora serrata. Therefore, the PAR (peripheral avascular retina) is defined as the nonperfusion area with measurements ≥ 2.0 DD, which is 3 standard deviations more than the normal value. Infants with persistent avascular retina have unknown long-term structural and functional risks, and theoretically could develop disease requiring treatment, including retinal breaks or tractional bands. Prolonged retinal traction by remnant shunt or extra-retinal fibrovascular proliferation between a stable prenatally vascularized retina in the posterior pole and an unstable postnatally vascularized retina may lead to the development of retinal holes characteristically located in the fragile, anterior undifferentiated avascular retina. Treatment options may vary from observation to retinal laser photocoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent peripheral avascular retina attending follow up till the age of 18 months in the core study whether;
* regressed ROP: children with regressed ROP who had not received any treatment.
* IVI treatment ROP: children with a history of threshold ROP treated with IVI of anti-VEGF agents.

Exclusion Criteria:

* Eyes with previous laser therapy.
* Eyes with any other pathology, other than ROP.
* Eyes with stage 4 or 5 ROP.
* Patients with hypersensitivity to iodinated contrast media, liver and renal insufficiency, history of asthma.
* Patients who will show hypersensitivity reaction to fluorescein angiography will be excluded from the thesis.
* Patients unfit for general anesthesia.

Ages: 18 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of eyes showing peripheral retinal active leakage. | 18 months
  Management of active leakage by laser ablation.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsai AS, Chou HD, Ling XC, Al-Khaled T, Valikodath N, Cole E, Yap VL, Chiang MF, Chan RVP, Wu WC. Assessment and management of retinopathy of prematurity in the era of anti-vascular endothelial growth factor (VEGF). Prog Retin Eye Res. 2022 May;88:101018. doi: 10.1016/j.preteyeres.2021.101018. Epub 2021 Nov 9. PMID 34763060
- [Result] Hellstrom A, Smith LE, Dammann O. Retinopathy of prematurity. Lancet. 2013 Oct 26;382(9902):1445-57. doi: 10.1016/S0140-6736(13)60178-6. Epub 2013 Jun 17. PMID 23782686
- [Result] Reynolds JD, Dobson V, Quinn GE, Fielder AR, Palmer EA, Saunders RA, Hardy RJ, Phelps DL, Baker JD, Trese MT, Schaffer D, Tung B; CRYO-ROP and LIGHT-ROP Cooperative Study Groups. Evidence-based screening criteria for retinopathy of prematurity: natural history data from the CRYO-ROP and LIGHT-ROP studies. Arch Ophthalmol. 2002 Nov;120(11):1470-6. doi: 10.1001/archopht.120.11.1470. PMID 12427059
- [Result] Mansukhani SA, Hutchinson AK, Neustein R, Schertzer J, Allen JC, Hubbard GB. Fluorescein Angiography in Retinopathy of Prematurity: Comparison of Infants Treated with Bevacizumab to Those with Spontaneous Regression. Ophthalmol Retina. 2019 May;3(5):436-443. doi: 10.1016/j.oret.2019.01.016. Epub 2019 Jan 31. PMID 31044736
- [Result] Klufas MA, Patel SN, Ryan MC, Patel Gupta M, Jonas KE, Ostmo S, Martinez-Castellanos MA, Berrocal AM, Chiang MF, Chan RV. Influence of Fluorescein Angiography on the Diagnosis and Management of Retinopathy of Prematurity. Ophthalmology. 2015 Aug;122(8):1601-8. doi: 10.1016/j.ophtha.2015.04.023. Epub 2015 May 28. PMID 26028345
- [Result] Lepore D, Quinn GE, Molle F, Orazi L, Baldascino A, Ji MH, Sammartino M, Sbaraglia F, Ricci D, Mercuri E. Follow-up to Age 4 Years of Treatment of Type 1 Retinopathy of Prematurity Intravitreal Bevacizumab Injection versus Laser: Fluorescein Angiographic Findings. Ophthalmology. 2018 Feb;125(2):218-226. doi: 10.1016/j.ophtha.2017.08.005. Epub 2017 Sep 1. PMID 28867130